CLINICAL TRIAL: NCT03671135
Title: A Prospective Multicenter Clinical Study to Evaluate the Safety and Effectiveness of Intrastromal Implant of the Transform Corneal Allograft (TCA) for Providing Near Vision in Presbyopic Subjects
Brief Title: Safety and Efficacy of an Intrastromal Transform™ Corneal Allograft (TCA) for Presbyopia Correction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Allotex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO_010
Record Dates: First submitted 2018-09-06; First posted 2018-09-14 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Presbyopia
Keywords: Intrastromal; Corneal Inlay
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCA Intrastromal Inlay (Experimental): A monocular intrastromal corneal inlay will be implanted.
  Interventions: Other: TCA Intrastromal Inlay

INTERVENTIONS:
Other: TCA Intrastromal Inlay — Anterior surface of Bowmans Layer Corneal Optical Correction Inlay

SUMMARY:
The objective of this clinical study is to evaluate the safety and effectiveness of intrastromal implantation of the Allotex TransForm corneal allograft (TCA) for improving near vision in presbyopic subjects.

DETAILED DESCRIPTION:
Beginning in 1949 with the pioneering work of Jose Barraquer, there has been an interest in using natural corneal tissue to change the refractive properties of the eye. In recent years, non-allogenic, synthetic corneal implants have received marketing approval in the United Stated and Europe for refractive purposes. Although synthetic implants are made of biocompatible materials they are not equivalent to an allogenic implant in terms of biocompatibility. The Allotex TCA is a piece of acellular cornea, sterilized with electron beam radiation and shaped to a particular shape using a laser. The availability of precise laser shaping systems and sterile corneas are the key factors that make the use of allogenic implants possible.

The TCA is placed in an intrastromal flap (Just beneath Bowmans layer) created using a femtosecond laser. The goal is to enhance the visual performance of the patient with a material that is 100% biocompatible and precisely shaped for the individual's needs.

Subjects must be presbyopic adults, needing from +1.75 D to +3.50 D of reading add in the non-dominant eye and must have uncorrected near visual acuity worse than 20/40 in the non-dominant eye. Bilateral treatments will not be allowed during this study.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent, have signed the written informed consent form, and been given a copy.
* Presbyopic adults, needing from +1.75 D to +3.50 D of reading add in the nondominant eye to improve near visual acuity at 40 cm by at least one line or more.
* Uncorrected near visual acuity worse than 20/40 in the non-dominant eye.
* Distance visual acuity correctable to at least 20/20 in both eyes.
* Near visual acuity correctable to at least 20/20 in both eyes.
* Manifest refraction spherical equivalent (MRSE) between -0.75 and +1.00 D with ≤0.75 D of refractive cylinder in the non-dominant eye.
* Stable vision, i.e. MSRE within 0.50 D over prior 12 months in the non-dominant eye.
* Contact lens wearers must discontinue hard or rigid gas permeable lenses for at least 2 weeks and discontinue soft lenses for at least 3 days prior to baseline examination.
* Contact lens wearers must have two (2) central keratometry readings with regular mires and two (2) manifest refractions taken at least one week apart, with no contact lens wear between. Keratometric values must not differ by more than ±0.50 D in any meridian and MRSE values must not differ more than ±0.50 D in the non-dominant eye.
* Average corneal power of ≥ 35.00 D and ≤ 47.00 D in the non-dominant eye.
* Subjects must be willing and able to return for scheduled follow-up examinations for 24 months after surgery.

Exclusion Criteria:

* A difference of > 0.75 D between the manifest refraction spherical equivalent and the cycloplegic refraction spherical equivalent in the non-dominant eye.
* Anterior segment pathology in the non-dominant eye.
* Signs or symptoms of clinically significant cataracts in the non-dominant eye.
* Residual, recurrent, active ocular or uncontrolled eyelid disease, or any corneal abnormality (including endothelial dystrophy, recurrent corneal erosion, etc.) in the non-dominant eye.
* Topographic signs of keratoconus (or keratoconus suspect) or other ectatic disorders in either eye.
* Subjects with clinically significant dry eyes, as determined by Tear Breakup Time (TBUT) of < 7 seconds or the presence of greater than mild symptoms of dryness or discomfort or SPK greater than grade 1.
* Distorted or unclear corneal mires on topography maps of the non-dominant eye.
* Macular degeneration, retinal detachment, or any other fundus pathology that would prevent an acceptable visual outcome in the non-dominant eye.
* Central corneal thickness <470 microns in either eye.
* Any prior intraocular surgery except corneal refractive surgery is allowed if performed more than 6 months prior to study participation.
* History of herpes zoster or herpes simplex keratitis in the non-dominant eye.
* History of steroid-responsive rise in intraocular pressure (IOP), preoperative IOP >21 mm Hg, glaucoma, or are a glaucoma suspect in the non-dominant eye.
* Using systemic medications with significant ocular side effects.
* Pregnant, lactating, or planning to become pregnant during the course of the study.
* Known sensitivity to planned study concomitant medications.
* Participating in any ophthalmic drug or device clinical trial during the time of this clinical investigation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the accuracy and stability of Presbyopic refractive correction following intervention with the Transform™ Corneal Allograft Inlay. | 6 months
  The primary effectiveness endpoint is an improvement in uncorrected near visual acuity (at 40 cm) at 6 months post-operativelyto20/40 or better. The goal is that more than 65% of eyes should have an uncorrected near visual acuity (UCNVA) of 20/40 or better at 6 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Vance Thompson, MD, Study Director — Study Medical Monitor/Consultant
Locations (4):
- Medipolis Wilrijk, Antwerp, Boomsesteenweg 223, Belgium
- Wellington Eye Clinic, Dublin, Beacon Court Sandyford, Ireland
- United Kingdom (2):
  - Corneo Plastic Unit and Eye Bank Queen Victoria Hospital, East Grinstead
  - Centre for Sight, London